CLINICAL TRIAL: NCT04200963
Title: A Phase 1a/b, Open-Label, Dose-Escalation and Expansion Study of IK-175, an Oral Aryl Hydrocarbon Receptor (AHR) Inhibitor, as a Single Agent and in Combination With Nivolumab, a PD-1 Checkpoint Inhibitor in Patients With Locally Advanced or Metastatic Solid Tumors and Urothelial Carcinoma
Brief Title: A Phase 1a/b Study of IK-175 as a Single Agent and in Combination With Nivolumab in Patients With Locally Advanced or Metastatic Solid Tumors and Urothelial Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ikena Oncology (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IK175-001; KYN-175 (Other: Ikena Oncology)
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Urothelial Carcinoma; Urothelial Carcinoma Bladder; Bladder Cancer; Bladder Disease; Solid Tumor; Solid Carcinoma; Solid Tumor, Adult; Metastatic Cancer; Advanced Solid Tumor; Advanced Cancer; Metastatic Bladder Cancer; Metastatic Urothelial Carcinoma; Locally Advanced Solid Tumor; Neoplasms; Neoplasm Metastasis; Neoplasm Malignant; Neoplasm, Bladder; Urothelial Neoplasm; Neoplasm, Urinary Bladder; Bladder Neoplasm; Bladder Urothelial Carcinoma
Keywords: IK-175; KYN-175; Immunoncology; Aryl Hydrocarbon Receptor Inhibitor; AHRi; Aryl Hydrocarbon Receptor Antagonist; Antagonist; Inhibitor; anti-PD1; nivolumab; checkpoint inhibitor; CPI; aPDI
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Urinary Bladder Diseases; Neoplasm Metastasis; Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion using the revised modified Toxicity Probability Interval (mTPI-2) design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- IK-175 Single Agent Dose Escalation (Experimental): Approximately 5 dose escalation steps are planned during the Single Agent Treatment dose escalation phase of the study. (COMPLETE)
  Interventions: Drug: IK-175
- IK-175 Single Agent Dose Expansion (Experimental): A Single Agent Treatment dose expansion phase will be performed in patients with urothelial carcinoma with IK-175 after completion of the dose escalation to confirm the RP2D. (COMPLETE)
  Interventions: Drug: IK-175
- IK-175 and nivolumab Combination Dose Escalation (Experimental): Approximately 2 dose escalation steps are planned during the Combination Treatment dose escalation phase of the study. (COMPLETE)
  Interventions: Drug: IK-175 and nivolumab
- IK-175 and nivolumab Combination Dose Expansion (Experimental): A Combination Treatment dose expansion phase will be performed in patients with urothelial carcinoma with IK-175 after completion of the dose escalation to confirm the RP2D. (COMPLETE)
  Interventions: Drug: IK-175 and nivolumab

INTERVENTIONS:
Drug: IK-175 — Subjects will be administered IK-175 PO daily for every 21-day treatment cycle during the Single Agent Treatment dose escalation or for every 28-day treatment cycle during the Single Agent dose expansion.
  Other Names: KYN-175
  Arms: IK-175 Single Agent Dose Escalation; IK-175 Single Agent Dose Expansion
Drug: IK-175 and nivolumab — Subjects will be administered IK-175 PO daily and administered a single dose of nivolumab IV on Day 1 for every 28-day treatment cycle during the Combination Treatment dose escalation and expansion.
  Other Names: KYN-175 and nivolumab
  Arms: IK-175 and nivolumab Combination Dose Escalation; IK-175 and nivolumab Combination Dose Expansion

SUMMARY:
This study will be conducted in adult subjects diagnosed with any form of an advanced or metastatic solid tumors including urothelial carcinoma for which standard therapy is no longer effective or is intolerable. This is a phase 1, multi-center, open label study designed to assess safety and tolerability of IK-175 as a single agent and in combination with nivolumab, to determine the recommended phase 2 dose (RP2D). Disease response, pharmacokinetics (PK), pharmacodynamics, and response biomarkers will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥18 years of age.
2. Patients with confirmed solid tumors (including urothelial carcinoma) who have locally recurrent or metastatic disease that has progressed on or following all standard of care therapies or who is not a candidate for standard treatment.
3. For patients with urothelial carcinoma to be enrolled in the Combination Treatment arm, patients must have confirmation of urothelial carcinoma and have unresectable locally recurrent or metastatic disease that has progressed on or following all standard of care therapies, or who is not a candidate for standard treatment. Checkpoint inhibitor therapy with anti-PD-1 or anti-PD-L1 does not necessarily need to directly precede the study, but patients must have progressed on or within 3 months of receiving the last infusion/dose anti-PD-(L)1 therapy for inclusion in the Combination Treatment arm only.
4. Have measurable disease.
5. Accessible tumor that can be safely accessed for multiple core biopsies and patient is willing to provide tissue from newly obtain biopsies before and during treatment.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
7. Adequate organ function.
8. Highly effective birth control.
9. Time since the last dose of prior therapy to treat underlying malignancy (including other investigational therapy): 9a. Systemic cytotoxic chemotherapy: ≥ the duration of the most recent cycle of the previous regimen (with a minimum of 2 weeks for all, except 6 weeks for systemic nitrosourea or systemic mitomycin-C). 9b. Biologic therapy (eg, antibodies): ≥ 3 weeks or their dosing interval if shorter than 3 weeks (e.g. q2w therapy would require a 2-week washout). 9c. Small molecule therapies: ≥ 5 × half-life. 9d. Investigational Agent: ≥4 weeks or ≥5 × half-life, whichever is shorter

Exclusion Criteria:

1. Untreated symptomatic central nervous system (CNS) tumors or brain metastasis. Patients are eligible if CNS metastases are asymptomatic and do not require immediate treatment or have been treated and patients have neurologically returned to baseline (residual signs or symptoms related to the CNS treatment are permitted). In addition, patients must have been either off corticosteroids, or on a stable or decreasing dose of ≤10 mg daily prednisone (or equivalent) for at least 2 weeks prior to entering the Treatment period (Day 1).
2. Patients who have not recovered to ≤ Grade 1 or baseline from all adverse events (AEs) due to previous therapies
3. Has an active autoimmune disease that has required systemic treatment in past 2 years with the use of disease-modifying agents, corticosteroids, or immunosuppressive drugs; nonsteroidal anti-inflammatory drugs (NSAIDs) are permitted. Patients with type 1 diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
4. Any condition requiring continuous systemic treatment with either corticosteroids (>10mg daily prednisone equivalents) or other immunosuppressive medications within 2 weeks prior to first dose of study treatment (Inhaled or topical steroids and physiological replacement doses of up to 10 mg daily prednisone equivalent are permitted in the absence of active clinically significant [ie, severe] autoimmune disease.).
5. Any other concurrent antineoplastic treatment or investigational agent except for allowed local radiation of lesions for palliation and hormone ablation.
6. Uncontrolled or life-threatening symptomatic concomitant disease (including known symptomatic human immunodeficiency virus (HIV) positive with an AIDS defining opportunistic infection within the last year, or a current CD4 count <350 cells/uL, symptomatic active hepatitis B or C checked at screening, or active tuberculosis). Patients with HIV are eligible if: 6a. they have received antiretroviral therapy (ART) for at least 4 weeks prior to entering the Treatment period as clinical indicated while enrolled on study; 6b. they continue on ART as clinically indicated while enrolled on study; 6c. CD4 counts and viral load are monitored per standard of care by a local health care provider.
7. Patients that have undergone a major surgery within 3 weeks of starting trial treatment or has inadequate healing or recovery from complications of surgery prior to starting trial treatment.
8. Prior radiotherapy within 2 weeks of start of study treatment. Subjects must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had severe radiation pneumonitis. A 1-week washout is permitted for palliative radiation [≤ 2 weeks of radiotherapy] to non-CNS disease.
9. Prior AHR inhibitor treatment without Sponsor permission.
10. Potentially life-threatening second malignancy requiring systemic treatment within the last 3 years or which would impede evaluation of treatment response. Hormone ablation therapy is allowed within the last 3 years. Patients with history of prior early stage basal/squamous cell skin cancer or non-invasive or in situ cancers that have undergone definitive treatment at any time are eligible.
11. Recent or current significant cardiovascular disease (e.g. stroke, heart attack, heart failure, or arrhythmia).
12. Medical issue that limits oral ingestion or impairment of gastrointestinal function that is expected to significantly reduce the absorption of IK-175.
13. Clinically significant (ie, active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or the presence of any condition that can increase proarrhythmic risk (eg, hypokalemia, bradycardia, heart block) including any new, unstable, or serious cardiac arrhythmia requiring medication, or other baseline arrhythmia that might interfere with interpretation of ECGs on study (eg, bundle branch block). Patients with QTcF >450 msec for males and >470 msec for females on screening ECG are excluded. Any patients with a bundle branch block will be excluded with QTcF >450 msec. Males who are on stable doses of concomitant medication with known prolongation of QTcF (eg, Selective Serotonin Reuptake Inhibitor Antidepressants) will only be excluded for QTcF >470 msec.
14. History of life-threatening toxicity related to prior immune therapy (eg. anti-CTLA-4 or anti-PD-1/PD-L1 treatment or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) except those that are unlikely to re-occur with standard countermeasures (eg. hormone replacement after adrenal crisis).
15. Has an active infection requiring systemic therapy.
16. Treatment with any live/attenuated vaccine within 30 days of first study treatment.
17. A woman of child-bearing potential (WOCBP) who has a positive pregnancy test or is breastfeeding prior to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated Dose (MTD) or Maximum Administered Dose (MAD), and to characterize the dose-limiting toxicities (DLTs) of IK-175 as a single agent and in combination with nivolumab. | Approximately 6 months
  Proportion of adverse events (AEs) meeting protocol-defined DLT criteria
Safety and tolerability of IK-175 as a single agent and in combination with nivolumab including acute and chronic toxicities, in determining a recommended phase 2 dose (RP2D) of IK- 175. | Up to 100 days after the end of study treatment.
  Frequency of AEs overall, by grade, relationship to study treatment, time-of-onset, duration of the event, duration of resolution, and concomitant medications administered.

SECONDARY OUTCOMES:
Pharmacokinetics of IK-175: half-life (t1/2) | Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 42 days) through end of treatment (average of 4 months)
  Determine IK-175 half-life (t1/2).
Pharmacokinetics of IK-175: Maximum Serum Concentration (Cmax) | Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 42 days) through end of treatment (average of 4 months)
  Determine IK-175 Cmax
Pharmacokinetics of IK-175: Area Under the Curve (AUC) | Days 1 and 2 of first 2 cycles (every 21 days), followed by Day 1 of every even cycle beginning with cycle 4 (every 42 days) through end of treatment (average of 4 months)
  Determine IK-175 AUC
Objective response rate (ORR) of IK-175 as a single agent and in combination with nivolumab | 12 months
  Preliminary antitumor activity per RECIST 1.1 and assessment per immune Response Evaluation Criteria Solid Tumors (iRECIST) for subjects with urothelial carcinoma.
Progression-free survival (PFS) of IK-175 as a single agent and in combination with nivolumab | 12 months
  Preliminary antitumor activity per RECIST 1.1and assessment per immune Response Evaluation Criteria Solid Tumors (iRECIST) for subjects with urothelial carcinoma.
Duration of treatment (DOT) of IK-175 as a single agent and in combination with nivolumab | 12 months
  Preliminary antitumor activity per RECIST 1.1 and assessment per immune Response Evaluation Criteria Solid Tumors (iRECIST) for subjects with urothelial carcinoma.
Duration of response (DOR) of IK-175 as a single agent and in combination with nivolumab | 12 months
  Preliminary antitumor activity per RECIST 1.1 and assessment per immune Response Evaluation Criteria Solid Tumors (iRECIST) for subjects with urothelial carcinoma.
Disease control rate (DCR) of IK-175 as a single agent and in combination with nivolumab | 12 months
  Preliminary antitumor activity per RECIST 1.1 and assessment per immune Response Evaluation Criteria Solid Tumors (iRECIST) for subjects with urothelial carcinoma.
Pharmacodynamic immune effects of IK-175 as a single agent and in combination with nivolumab on tumor-infiltrating cytotoxic T cells | Prior to Cycle 1 Day 1, and anytime between the end of Cycle 1 and end of Cycle 2. Each cycle is 21 days.
  Characterization of tumor-infiltrating cytotoxic T cells in tumor biopsies collected before and during IK-175 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Karim Malek, MD, Study Director — Ikena Oncology
Locations (10):
- United States (10):
  - Banner Health- MD Anderson Cancer Center, Gilbert, Arizona
  - Florida Cancer Specialists - Sarasota, Sarasota, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Johns Hopkins Kimmel Cancer Center, Baltimore, Maryland
  - START Midwest, Grand Rapids, Michigan
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Sydney Kimmel Cancer Center Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No